CLINICAL TRIAL: NCT06241469
Title: Efficacy and Safety of Sintilimab Combined With Nab-paclitaxel and Tegio (aTS) as First-line Treatment of Unresectable Locally Advanced, Recurrent or Metastatic Adenocarcinoma of Gastric and Gastroesophageal Junction (CZTU-1)：a Phase II Clinical Study
Brief Title: Efficacy and Safety of Sintilimab Combined With Nab-paclitaxel and Tegio (aTS) as First-line Treatment of Unresectable Locally Advanced, Recurrent or Metastatic Adenocarcinoma of Gastric and Gastroesophageal Junction，a Phase II Clinical Study
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wu Jun (Other)
Responsible Party: Sponsor-Investigator, Wu Jun, Professor, The First People's Hospital of Changzhou
Organization: The First People's Hospital of Changzhou (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMCC201312
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Gastric Cancer; GastroEsophageal Cancer; Adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms; Adenocarcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): Sintilimab combined with nab-paclitaxel and tegio
  Interventions: Drug: Sintilimab,nab-paclitaxel and tegio

INTERVENTIONS:
Drug: Sintilimab,nab-paclitaxel and tegio — Immunotherapy combined with chemotherapy

SUMMARY:
The goal of this clinical trial is to find better protocal for adenocarcinoma of the gastric and gastroesophageal juncion.

The main question is aim to answer is:

1. The efficacy and safety of PD-1 monoclonal antibody (Sintilimab) combined with nab-paclitaxel and S-1 in the first-line treatment of advanced gastric and gastroesophageal junction adenocarcinoma.

Participants will be given PD-1 monoclonal antibody, nab-paclitaxel and tegio.

ELIGIBILITY:
Inclusion Criteria:

1. Non resectable locally advanced, recurrent, or metastatic adenocarcinoma at the junction of the stomach and esophagus (including signet ring cell carcinoma, mucinous adenocarcinoma, and hepatoid adenocarcinoma) confirmed by histopathological examination.
2. Age ≥ 18 years old.
3. The ECOG PS score is 0 or 1.
4. The time from the end of previous (new) adjuvant chemotherapy/radiotherapy to disease recurrence is greater than 6 months.
5. Palliative treatment for local lesions (non target lesions) should last for more than 2 weeks until randomization.
6. According to RECIST v1.1, there should be at least one measurable or evaluable lesion.
7. Can provide archived or fresh pathological tissues within 6 months from the signing of the informed consent document for PD-L1 testing and obtain test results.
8. Having sufficient organ and bone marrow functions, defined as follows:

1) Blood routine: Absolute neutrophil count (ANC) ≥ 1.5 × 109/L; Platelet count (PLT)≥ 100 × 109/L; Hemoglobin content (HGB) ≥ 8.0 g/dL. No G-CSF, GM-CSF, Meg CSF, TPO, EPO, red blood cell transfusions or platelet transfusions were not used within the first 7 days of the examination.

2) Liver function: Patients without liver metastasis require serum total bilirubin (TBIL) ≤ 1.5 × Normal upper limit (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN. Patients with liver metastasis require serum total bilirubin (TBIL) ≤ 1.5 × Normal upper limit (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 × ULN.

3) Renal function: Glomerular filtration rate (GFR) ≥ 60 mL/min(Calculate using the CKD-EPI formula) 4) Adequate coagulation function is defined as an international standardized ratio (INR) ≤ 1.5 or prothrombin time (PT) ≤ 1.5 × ULN; If the subject is receiving anticoagulant treatment, as long as the PT is within the range of anticoagulant drugs prescribed; 5) Urinary routine: Urinary protein<2+; If the urine protein is ≥ 2+, the 24-hour urine protein quantification needs to be<1.0 g.

9. Expected survival time ≥ 24 weeks. 10. Female participants of childbearing age or male participants whose sexual partners are female participants of childbearing age are required to take effective contraceptive measures throughout the entire treatment period and 6 months after the treatment period.

11. Sign a written informed consent form and be able to comply with the visitation and related procedures stipulated in the plan.

Exclusion Criteria:

1. Known signs of active bleeding in the lesion (excluding positive fecal occult blood).
2. Obstruction of the cardia and pylorus can affect the patient's eating and gastric emptying, or hinder the swallowing of medication.
3. Diagnosed as HER2 positive adenocarcinoma at the junction of the stomach and esophagus.
4. Previously received systematic treatment for advanced or metastatic adenocarcinoma at the junction of the stomach and esophagus.
5. Peripheral neurotoxicity has not recovered to level 1 after previous treatment.
6. It is known that dihydropyrimidine dehydrogenase (DPD) is deficient (or has experienced mucosal toxicity of grade 3 or higher in previous fluorouracil containing treatments).
7. Known to be allergic to any monoclonal antibody or chemotherapy drug (tigio, albumin bound paclitaxel) formulation component (having experienced grade 3 or above allergic reactions).
8. Previously exposed to any anti-PD-1 or anti-PD-L1, PD-L2, CD137, CTLA-4 antibody therapy, or any other antibody or drug targeting T cell co stimulation or checkpoint pathways.
9. Participate in another intervention clinical study at the same time, unless participating in an observational (non intervention) clinical study or in the follow-up stage of an intervention study.
10. Within 2 weeks before the first administration, systemic systemic treatment with Chinese herbal medicine or immunomodulatory drugs (including thymosin, interferon, interleukin, etc.) with anti-tumor indications has been received;
11. Within 4 weeks prior to the first dose of study treatment, immunosuppressive drugs were used, excluding local corticosteroids administered through nasal spray, inhalation, or other routes, or systemic corticosteroids administered at physiological doses (i.e. no more than 10 mg/day of prednisone or equivalent doses of other corticosteroids), or steroids were used to prevent contrast agent allergies.
12. Within 4 weeks prior to the first dose of study treatment or planned to receive attenuated live vaccines during the study period.

    Note: It is allowed to receive inactivated viral vaccines for seasonal influenza within 4 weeks before the first administration; But it is not allowed to receive attenuated live influenza vaccines;
13. Have undergone major surgical procedures (craniotomy, thoracotomy, or laparotomy) within 4 weeks prior to the first dose of study treatment, or are expected to require major surgery during the study treatment period; Laparoscopic exploration surgery was performed within 2 weeks prior to the first dose of study treatment.
14. Toxicity (excluding hair loss, non clinically significant, and asymptomatic laboratory abnormalities) at level 0 or 1 of the National Cancer Institute Common Standard Terminology 5.0 (NCI CTCAE v5.0) caused by previous anti-tumor treatments prior to the initial study treatment.
15. It is known that there are symptomatic central nervous system metastases and/or cancerous meningitis. For subjects with brain metastases who have received previous treatment, if their condition is stable (no evidence of imaging progression at least 4 weeks prior to the first administration of the trial treatment, and repeated imaging examinations confirm no evidence of new or enlarged brain metastases), and they do not require steroid treatment for at least 14 days prior to the first administration of the trial treatment, they can participate in the trial. This exception does not include cancerous meningitis, which should be excluded regardless of its stable clinical condition.
16. Any ascites that can be detected during physical examination, ascites that have been previously treated or still require treatment, with only a small amount of ascites shown on imaging but no symptoms, can be selected.
17. Patients with equal amount of fluid accumulation in both sides of the chest cavity, or a large amount of fluid accumulation in one side of the chest cavity, or those who have caused respiratory dysfunction and require drainage.
18. Patients with bone metastases who are at risk of paralysis.
19. Known or suspected autoimmune disease or medical history of the disease in the past two years (vitiligo, psoriasis, alopecia or Grave's disease that does not need systematic treatment in the past two years, hypothyroidism that only needs thyroid hormone replacement therapy and type I diabetes patients that only need insulin replacement therapy can be included in the group).
20. Known history of primary immunodeficiency.
21. Known to have active pulmonary tuberculosis.
22. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
23. Known history of human immunodeficiency virus (HIV) infection (i.e. HIV antibody positive).
24. Severe infections that are active or poorly controlled clinically.
25. Symptomatic congestive heart failure (New York Heart Association classification II-IV) or symptomatic or poorly controlled arrhythmia.
26. Uncontrolled arterial hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg) even after receiving standardized treatment.
27. Have experienced any arterial thromboembolism events, including myocardial infarction, unstable angina, cerebrovascular accidents, or transient ischemic attacks, within the 6 months prior to enrollment for treatment.
28. Significant malnutrition (a weight loss of 5% within 1 month of signing the informed consent form, a weight loss of>15% within 3 months, or a decrease of 1/2 or more in food intake within 1 week), except for malnutrition correction of more than 4 weeks before the first dose of study drug administration.
29. A history of deep vein thrombosis, pulmonary embolism, or any other severe thromboembolism within the 3 months prior to enrollment (implantable venous infusion port or catheter-related thrombosis, or superficial venous thrombosis is not considered "severe" thromboembolism).
30. Uncontrolled metabolic disorders or other non malignant organ or systemic diseases or secondary reactions to cancer, which can lead to higher medical risk and/or uncertainty in survival evaluation.
31. Hepatoencephalopathy, hepatorenal syndrome, or Child Pugh B grade or more severe cirrhosis.
32. History of tumor related intestinal obstruction (within 3 months prior to the signing of informed consent) or the following diseases: inflammatory bowel disease or extensive bowel resection (partial or extensive bowel resection with concurrent chronic diarrhea), Crohn's disease, ulcerative colitis.
33. Known to have acute or chronic active hepatitis B virus (HBsAg positive and HBV DNA viral load ≥ 200 IU/mL or ≥ 103 copy number/mL) or acute or chronic active hepatitis C virus (HCV antibody positive and HCV RNA positive).
34. Active syphilis infected individuals who require treatment.
35. There is a history of gastrointestinal perforation and/or fistula within the 6 months prior to enrollment in the study, except for patients with gastric cancer perforation who have undergone surgical resection of the primary lesion of gastric cancer.
36. Suffering from interstitial lung disease that requires steroid hormone treatment.
37. History of other primary malignant tumors, excluding:

    * Complete remission (CR) of malignant tumors for at least 2 years prior to enrollment and no additional treatment required during the study period;
    * Non melanoma skin cancer or malignant freckle like nevi that have been adequately treated and have no evidence of disease recurrence;
    * In situ cancer with sufficient treatment and no evidence of disease recurrence.
38. Pregnant or breastfeeding female patients.
39. Other acute or chronic diseases, mental illnesses, or abnormal laboratory test values that may lead to increased risk of study participation or drug administration, or interference with the interpretation of study results, and the inclusion of patients as ineligible to participate in this study based on the researcher's judgment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-03 (Estimated); Primary Completion 2026-08-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | from randomization up to progressive disease or EOT due to any cause, assessed up to 2 year
  Tumor assessment will be performed using radiography method every 6 weeks, until the occurrence of progressive disease (PD), using RECIST v 1.1
Objective response rate (ORR) | from randomization up to progressive disease or EOT due to any cause, assessed up to 2 year
  Tumor assessment will be performed using radiography method every 6 weeks, until the occurrence of progressive disease (PD), using RECIST v 1.1

SECONDARY OUTCOMES:
Overall survival (OS) | from randomization up to progressive disease or EOT due to any cause, assessed up to 2 year
  Tumor assessment will be performed using radiography method every 6 weeks, until the occurrence of progressive disease (PD), using RECIST v 1.1
Disease control rate (DCR) | from randomization up to progressive disease or EOT due to any cause, assessed up to 2 year
  Tumor assessment will be performed using radiography method every 6 weeks, until the occurrence of progressive disease (PD), using RECIST v 1.1
Disease control rate (DOR) | from randomization up to progressive disease or EOT due to any cause, assessed up to 2 year
  Tumor assessment will be performed using radiography method every 6 weeks, until the occurrence of progressive disease (PD), using RECIST v 1.1

CONTACTS AND LOCATIONS:
Locations (1):
- The First People's Hospital of Changzhou, Changzhou, Jiangsu, China